CLINICAL TRIAL: NCT05211349
Title: Psychometric Evaluation of Dual-Task Timed Get Up and Go Test (Cognitive) and 3-m Backwards Back Test in Community-dwelling Stroke Individuals
Brief Title: Comparison of Dual-Task Timed Up and Go Test (Cognitive) and 3-m Backwards Walk Test
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Emel Taşvuran Horata, PhD; Assistant Professor, Afyonkarahisar Health Sciences University
Other Study IDs: 2021/534
Record Dates: First submitted 2022-01-23; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Stroke
Keywords: Stroke; Falling; Reliability and Validity; Postural Balance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Dual-Task Timed Up and Go Test (cognitive) — It evaluates balance with a simultaneous cognitive and motor task. The cognitive task of the test is serial triple subtraction while the TUG test is a motor task. Balance performance will be recorded in seconds.
Other: 3-m Backward Walk Test — It is used to assess fall risk and balance. It is calculated in how many seconds an individual can walk backward a marked distance of 3 meters.
Other: Modified Four Square Step Test — It is a performance test that evaluates dynamic balance in stroke individuals with the ability to avoid obstacles and take steps in all directions. Balance performance is recorded in seconds.
Other: Timed Up and Go Test — It is used to assess balance and functional mobility. The participant is asked to get up from the chair she/he is sitting in, walk the marked distance of 3 meters and return to her/his seat again. The elapsed time is recorded in seconds.
Other: Berg Balance Test — It consists of 14 items and evaluates dynamic balance and functional mobility in stroke. The maximum score is 56. Higher scores indicate better balance.

SUMMARY:
Two balance assessment tools that have been used recently have attracted considerable attention: the Dual-Task Timed Up and Go Test (cognitive) (DTUG) and the 3-m Backward Walk Test (3MBWT). The aim of this study is to compare the psychometric properties of two clinically proven balance assessment tools.

DETAILED DESCRIPTION:
There are unidimensional and multidimensional scales used to evaluate gait balance after stroke. Unidimensional scales (DTUG, 3MBWT) can be useful in clinical practice and in screening for basic balance problems. Two balance assessment tools that have been used recently have attracted considerable attention: the Dual-Task Timed Up and Go Test (cognitive) (DTUG) and the 3-m Backward Walk Test (3MBWT). The aim of this study is to compare the psychometric properties of two clinically proven balance assessment tools. In the study, construct validity, concurrent validity, reliability, and cut-off score (for determining falling risk) of the two tests will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Single stroke with unilateral hemiparesis at least 6 months prior to the study,
* Be in the age range of 50-85 years
* Able to walk at least 10 meters independently with or without a walking aid,
* Getting at least 24 points from the Standardized Mini-Mental Test
* It is to be able to follow two-stage commands and perform subtraction.

Exclusion Criteria:

* Presence of additional orthopedic or neurological diseases that may affect balance and walking,
* Having uncorrected vision and hearing problems

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All of the participants will consist of stroke individuals who receive inpatient or outpatient treatment in the Physical Therapy and Rehabilitation Polyclinic. All assessments will be done face to face. Men and women aged 50-85 years who have had a stroke for at least 6 months will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-01-02 (Actual); Primary Completion 2023-01-02 (Estimated); Study Completion 2024-01-02 (Estimated)

PRIMARY OUTCOMES:
Dual-Task Timed Up and Go Test (cognitive) | 5 minutes
  It evaluates balance and functional mobility with a simultaneous cognitive and motor task. The cognitive task of the test is 3-series subtraction, while the TUG test is the motor task. Performance is recorded in seconds.
3-m Backward Walk Test | 5 minutes
  It is used to assess fall risk and balance. It is calculated in how many seconds an individual can walk backwards a marked distance of 3 meters.

CONTACTS AND LOCATIONS:
Overall Officials: EMEL TAŞVURAN HORATA, PhD, Principal Investigator — AFSU
Locations (1):
- Afyonkarahisar Health Science University, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tasvuran Horata E, Eken F, Taskin G, Kara G, Yesil H, Adar S, Baskan E, Dundar U. Comparison of psychometric properties of the dual-task timed up-and-go test (cognitive) and the 3-m walk backward test in community-dwelling stroke patients. Top Stroke Rehabil. 2025 Mar;32(2):140-149. doi: 10.1080/10749357.2024.2377514. Epub 2024 Jul 14. PMID 39003753